CLINICAL TRIAL: NCT06240598
Title: Identification of Markers of Resistance During Frontline Therapy and Maintenance
Brief Title: A Study of Second Look Laparoscopy (SLL) in People With Ovarian Cancer Who Have Completed Their First Course of Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-249
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
Keywords: stage III-IV; epithelial ovarian cancer; second Look Laparoscopy (SLL); 23-249
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: This is a prospective study for biospecimen collection during standard of care procedures and during second look laparoscopy (SLL), which constitutes the only investigational procedure in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second Look Laparoscopy (SLL) (Experimental): Patients will be treated with standard of care observation or maintenance therapy as per investigator decision.The only investigational intervention performed through this study is the SLL.
  Interventions: Procedure: Second Look Laparoscopy

INTERVENTIONS:
Procedure: Second Look Laparoscopy — Second Look Laparoscopy (SLL)

SUMMARY:
The researchers are doing this study to look at the health outcomes of people with advanced ovarian cancer who have a second look laparoscopy (SLL) after they complete their first course of chemotherapy. The researchers will compare the health outcomes of people who have minimal residual disease (MRD-small amounts of cancer cells in the body after a person receives treatment) at the time of SLL with the health outcomes of people who do not have MRD at the time of SLL. The researchers are also doing this study to determine if SLL is safe and practical (feasible) in people with advanced ovarian cancer who have completed the first course of therapy for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned female at birth≥ 18 years of age
* Suspected or known stage III-IV epithelial ovarian cancer for which the patient has undergone, or is planned to undergo, attempted primary or interval debulking surgery
* Homologous Recombination Deficiency testing should be planned to be completed prior to completion of initial platinum/taxane chemotherapy. HRD testing can be determined using :

  * Confirmation of deleterious Somatic or Germline BRCA mutation
  * CLIA certified test for HRD
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or drainage gastrostomy tube
* Patients receiving standard of care or investigational protocol directed treatment are eligible for this study, with the exception of protocol directed treatment which would prohibit the SLL surgery from being performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer
Enrollment: 80 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
minimal residual disease (MRD) status | up to 12 weeks
  will be based on surgicopathological findings from multiple biopsies and peritoneal cytology obtained during the SLL procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grisham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk -Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm